CLINICAL TRIAL: NCT04896541
Title: A Phase I Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD7442 in Healthy Japanese Participants
Brief Title: Phase I Double-blind, Placebo-controlled Study of AZD7442
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D8850C00005; NCT05406375 (obsolete NCT alias)
Record Dates: First submitted 2021-02-26; First posted 2021-05-21 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD7442 (Experimental): Single dose (IM injections or IV administration) of AZD7442 or saline placebo on Day 1.
  Interventions: Biological: AZD7442 300 mg IM(male); Biological: AZD7442 600 mg IM (male); Biological: AZD7442 300 mg IV (male and female); Biological: AZD7442 1000 mg IV (male)
- placebo (Experimental): Single dose (× 2 separate IM injections or IV administration) of AZD7442 or saline placebo on Day 1.
  Interventions: Biological: AZD7442 300 mg IM(male); Biological: AZD7442 600 mg IM (male); Biological: AZD7442 300 mg IV (male and female); Biological: AZD7442 1000 mg IV (male)

INTERVENTIONS:
Biological: AZD7442 300 mg IM(male) — Single dose of 300 mg of AZD7442 or saline placebo on Day 1.
Biological: AZD7442 600 mg IM (male) — Single dose of 600 mg of AZD7442 or saline placebo on Day 1.
Biological: AZD7442 300 mg IV (male and female) — Single dose of 300 mg of AZD7442 or saline placebo on Day 1.
Biological: AZD7442 1000 mg IV (male) — Single dose 1000 mg of AZD7442 or saline placebo on Day 1.

SUMMARY:
AZD7442 mAbs are being evaluated for administration to prevent or treat COVID-19. This Phase I study will gather important information on the safety and tolerability of AZD7442.

DETAILED DESCRIPTION:
Severe acute respiratory coronavirus 2 is a novel coronavirus that appears to have first emerged in China in November 2019 causing cases of atypical pneumonia. Since then, the COVID-19 pandemic has caused major disruption to healthcare systems with significant socioeconomic impacts. As of 22 December 2020, the virus had spread to all corners of the globe, involving 218 countries/regions with over 78.00 million confirmed cases reported and more than 1.71 million associated deaths. As a response to the ongoing pandemic, AstraZeneca is developing mAbs to the SARS-CoV-2 spike protein. The SARS-CoV-2 spike protein contains the virus's receptor binding domain, which enables the virus to bind to receptors on human cells. By targeting this region of the virus's spike protein, antibodies can block the virus's attachment to human cells, and, therefore, are expected to block infection. AZD7442, a combination of 2 of these mAbs (AZD8895 and AZD1061), is being evaluated for administration to treat or prevent COVID-19. There are currently one ongoing Phase I study and two ongoing Phase III studies with AZD7442, in addition to this treatment study.

Randomization of approximately 40 Japanese participants is planned.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be Japanese men and women and 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Negative results from both SARS-CoV-2 qRT-PCR and serology tests
* Healthy by medical history, physical examination, and safety laboratory tests, according to the judgement of the investigators

Exclusion Criteria:

* Fever above 37.5°C by the time when the participant is randomised; a participant excluded for transient acute illness may be dosed if the illness resolves by the time of randomisation.
* History of infection with SARS or MERS
* Any drug therapy within 7 days prior to Day 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Adverse event and serious adverse event | Up to Day361
  To evaluate the safety and tolerability of AZD7442 administered IV or IM_Adverse event and serious adverse event
Pharmacokinetics - Serum Concentration | Up to Day361
  To evaluate the single-dose PK of AZD7442.
Pharmacokinetics - Maximum Serum Concentration | Up to Day361
  To evaluate the single-dose PK of AZD7442.
Pharmacokinetics - Time to Maximum Serum Concentration | Up to Day361
  To evaluate the single-dose PK of AZD7442.
Pharmacokinetics - Area under the plasma concentration-time curve to the last measurable time point | Up to Day361
  To evaluate the single-dose PK of AZD7442.
Pharmacokinetics - Area under the plasma concentration-time curve extrapolated to infinity | Up to Day361
  To evaluate the single-dose PK of AZD7442.
Pharmacokinetics - extravascular systemic clearance | Up to 361
  To evaluate the single-dose PK of AZD7442.
Pharmacokinetics -bioavailability | Up to Day361
  To evaluate the single-dose PK of AZD7442.
Pharmacokinetics -extravascular terminal phase volume of distribution | Up to Day361
  To evaluate the single-dose PK of AZD7442.

SECONDARY OUTCOMES:
The serum neutralizing responses against SARS-CoV-2 using Geometric mean fold rise from baseline | Up to Day361
  Blood samples as neutralizing responses against SARS-CoV-2 in serum will be collected.
ADA responses to the AZD7442 in serum. | Up to Day361
  Blood samples for determination of ADA in serum will be assayed by bioanalytical test sites, using an appropriately validated bioanalytical method.
The serum neutralizing responses against SARS-CoV-2 using Geometric mean titre from baseline | Up to Day361
  Blood samples as neutralizing responses against SARS-CoV-2 in serum will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indeed that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Okada H, Ishikawa K, Itoh Y, Noda Y, Eto T, Pilla Reddy V, Chen CC, Gibbs M, Johnsson E. Safety, tolerability, and pharmacokinetics of half-life extended SARS-CoV-2-neutralizing monoclonal antibodies AZD7442 (tixagevimab/cilgavimab) in healthy Japanese adults. J Infect Chemother. 2023 Nov;29(11):1061-1067. doi: 10.1016/j.jiac.2023.07.014. Epub 2023 Jul 29. PMID 37524201
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343